CLINICAL TRIAL: NCT06869070
Title: Optimisation and Standardization of Circulating Cell-free DNA Ex-traction Protocols in a Diagnostic Setting
Acronym: OPTICIRC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: OPTICIRC
Record Dates: First submitted 2025-02-07; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Short term
- Long term

SUMMARY:
comparison of blood collection tubes and cell-free DNA extraction to evaluate the best possible combination to obtain high quantity and quality cell-free DNA sample for NGS analyses

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* no serious condition

Exclusion Criteria:

* younger than 18 years
* serious health condition that leads to higher cfDNA content in blood

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population has to be older than 18 years, can be of any gender and have a disease-free status
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
cfDNA quantity | Baseline, at enrollment
  we will assess the quantities in ng/µl of cell-free DNA extracted from plasma
cfDNA quality | Baseline, at enrollment
  we will assess the fragments length in nucleotides using TermoFisher's Tapestation from the extracted plasma cell-free DNA